CLINICAL TRIAL: NCT01912365
Title: Splinting Versus Above Elbow Casting for Type I Supracondylar Fractures of the Humerus in Children: A Randomized Controlled Trial
Brief Title: Splinting Versus Casting for Type I Supracondylar Fractures
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principle Investigator, University of British Columbia
Other Study IDs: H13-01520
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Bone Fractures
Keywords: Fracture; Supracondylar; Pediatric; Orthopedic
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Above Elbow Cast + Collar/cuff: Participants randomized to this group will be treated with an Above Elbow Cast & collar/cuff for 3 weeks
  Interventions: Procedure: Above Elbow Cast
- Long Arms Splint + Collar/Cuff: Participants randomized to this group will be treated with a long arm splint & collar/cuff for 3 weeks
  Interventions: Procedure: Long Arm Splint

INTERVENTIONS:
Procedure: Above Elbow Cast
  Groups: Above Elbow Cast + Collar/cuff
Procedure: Long Arm Splint
  Groups: Long Arms Splint + Collar/Cuff

SUMMARY:
Elbow fractures are very common in young children. Type I supracondylar fractures are stable fractures to the elbow that are treated conservatively across the world and typically heal very well without complications. There are several treatment options, including an above elbow cast or long arm splint. This study aims to determine if one treatment is no worse than the other in order to standardize the treatment of these fractures at our institution. The investigators hope to save families from extra hospital visits and reduce the amount of x-rays required for treatment of these fractures.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-12
* Type 1 supracondylar fracture

Exclusion Criteria:

* A type 2 or 3 supracondylar fracture
* Neurovascular compromise associated with the fracture
* Previous diagnosis with a metabolic or structural bone disease
* Other fractures to ipsilateral upper extremity
* History of injury to affected elbow

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible participants will be recruited from the Emergency Department at BC Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Baumann's Angle | 6 Months
  Baumann's angle of the injured elbow will be measured 6 months following the injury

SECONDARY OUTCOMES:
Humero-Capitellar Angle | 6 Months
  Humero-Capitellar Angle will be measured 6 Months following the injury
Functional Outcome Questionnaire | 6 Months
  All participants will complete the Activity Scale for Kids-P 6 months following the injury

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, MBBS, MS, MHSc, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Siu C, Farrell S, Schaeffer EK, Doan Q, Dobbe A, Bone J, Reilly CW, Mulpuri K. Long-Arm Splinting Versus Above-Elbow Casting for Type 1 Supracondylar Fractures of the Humerus in Children: a Randomized Controlled Trial. SN Compr Clin Med. 2023;5(1):72. doi: 10.1007/s42399-023-01417-z. Epub 2023 Feb 3. PMID 36776416